CLINICAL TRIAL: NCT00844220
Title: Coronary Artery Disease Management Using Multislice Computed Tomography and Magnetic Resonance Imaging
Acronym: CAD-Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Muenster (Other); Charite University, Berlin, Eva Schönenberger, MD (Unknown); University of Freiburg (Other)
Responsible Party: Principal Investigator, Marc Dewey, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EA1/080/08
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: Suspected coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Catheterization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT/MR (Experimental): CT/MRI-directed clinical management strategy
  Interventions: Procedure: CT/MR
- Catheterization (Active Comparator): Standard clinical management
  Interventions: Procedure: Catheterization

INTERVENTIONS:
Procedure: CT/MR — CT/MRI-directed clinical management strategy
  Arms: CT/MR
Procedure: Catheterization — Standard clinical management directed by conventional coronary angiography
  Arms: Catheterization

SUMMARY:
The primary objective of this study is to analyze the clinical value of a therapeutic management strategy based on the results of coronary CT angiography and functional MRI. The clinical value of CT and MRI will be analyzed in patients with suspected coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Suspected coronary artery disease and planned conventional coronary angiography based on atypical angina pectoris

Exclusion Criteria:

* Known coronary artery disease
* ST elevation
* Age below 30 years
* Women of child-bearing potential without a negative pregnancy test
* Inclusion in another study
* Heart rate above 70 beats per min and contraindications to beta blockers
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block
* Inability to hold the breath for 10 s

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2009-02-18 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Complications | during or up to 2 days after procedures
  Death, stroke, and myocardial infarction and moderate to severe groin hematoma, groin pain, infections, allergies, thromboses, and arteriovenous fistula or other complications (if prolonging the in-hospital stay significantly by at least 24 hours).

SECONDARY OUTCOMES:
Hard Cardiovascular Events | Follow-up 3 (36-60 Months)
  Composite endpoint: The most important secondary outcome will be hard cardiovascular events at final follow-up (3 years). These hard events include: cardiac and noncardiac death (death from any cause), stroke, and myocardial infarction. These hard events are considered as major adverse cardiovascular events.
Comparison of Contrast Induced Nephropathy | Follow-up 1 (6-12 Months), Follow-up 2 (12-24 Months), Follow-up 3 (36-60 Months)
  To compare contrast-induced nephropathy (CIN) defined as increase in creatinine by 25% or 0.5 mg/dl from baseline at the measurements obtained 18 to 24 and/or 46 to 50 hours after the initial procedures as part of standard safety parameters performed at our institution. In addition, CIN will also be assessed during the follow-ups.
Comparison of Comparison of Soft Cardiovascular Events | Follow-up 3 (36-60, Months)
  To compare soft cardiovascular events (unstable angina pectoris, re-revascularization, and first revascularization at least 2 months after randomization, according to the results of Ladenheim et al. J Am Coll Cardiol 1986, at final follow-up.
Comparison of In-Hospital Stay | Up to 24 hours after the end of the in-hospital stay.
  to compare the in-hospital stay time and overall length of stay.
Quality of Life Analysis | Follow-up 1 (6-12 Months), Follow-up 2 (12-24 Months), Follow-up 3 (36-60 Months)
  To analyze the change in quality of life (QALY) in both groups (prior to the tests and at follow-up) using the SF-12 and the EuroQuol as general measurement tools and the MacNew questionnaire as disease-specific questionnaire.
Confounding Effects of Nutrition, Physical Activity, and Depression | Follow-up 1 (6-12 Months), Follow-up 2 (12-24 Months), Follow-up 3 (36-60 Months)
  To analyze the effect and potentially confounding effect of nutrition, physical activity (using the Freiburg questionnaire), and depression (assessed with the HADS questionnaire) in the two groups.
Comparison of Cost-effectiveness | Follow-up 3 (36-60 Months)
  To compare cost-effectiveness in both groups using the primary and secondary efficacy data, the QALY data, and cost data derived from the trial.
Comparison of Patient Preference | 24 hours after last procedure related to computed tomography or conventional coronary angiography
  To analyze patient preference and satisfaction with the therapeutic management strategies with a focus on the comfort during the imaging tests.
Comparison of the Amount of Contrast Agent | 10 minutes after the examinations.
  Comparison of the amount of contrast agent
Comparison of the Amount of Radiation Exposure | Comparison of the amount of radiation exposure
  10 minutes after computed tomography or conventional coronary angiography
Analysis of Image Quality | Up to 24 hours after the end of computed tomography
  To analyze which image quality in multislice computed coronary angiography would be required to directly reliably triage patients to coronary artery bypass grafting.
Analysis of Correlation and Agreement About the Stenosis Diameter Between Multislice Computed Coronary Angiography and Conventional Coronary Angiography | Up to 24 hours after the end of computed tomography
  To analyze the correlation and agreement between multislice computed coronary angiography and conventional coronary angiography (using quantitative analysis) for estimation of the percent diameter stenosis in patients who underwent both tests.
Comparison of Biological Effects of Radiation Exposure | Z1) before exam, (Z2) 60 min after end of exam, (Z3) 18-24h after exam
  To compare the biological effects of radiation exposure of ionizing radiation, measured by DNA double-strand breaks in lymphocytes, of CT and conventional coronary angiography themselves and in the two randomization groups (approval by ethics board for this substudy with start of first patient analyzed on September, 15, 2009). Blood samples are taken for double-strand break analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- [Background] Dewey M, de Vries H, de Vries L, Haas D, Leidecker C. The present and future of cardiac CT in research and clinical practice: moderated discussion and scientific debate with representatives from the four main vendors. Rofo. 2010 Apr;182(4):313-21. doi: 10.1055/s-0029-1245195. Epub 2010 Mar 16. PMID 20234975
- [Background] Zimmermann E, Dewey M. Whole-heart 320-row computed tomography: reduction of radiation dose via prior coronary calcium scanning. Rofo. 2011 Jan;183(1):54-9. doi: 10.1055/s-0029-1245629. Epub 2010 Aug 19. PMID 20725881
- [Background] Dewey M, Zimmermann E, Deissenrieder F, Laule M, Dubel HP, Schlattmann P, Knebel F, Rutsch W, Hamm B. Noninvasive coronary angiography by 320-row computed tomography with lower radiation exposure and maintained diagnostic accuracy: comparison of results with cardiac catheterization in a head-to-head pilot investigation. Circulation. 2009 Sep 8;120(10):867-75. doi: 10.1161/CIRCULATIONAHA.109.859280. Epub 2009 Aug 24. PMID 19704093
- [Background] Dewey M. Coronary CT versus MR angiography: pro CT--the role of CT angiography. Radiology. 2011 Feb;258(2):329-39. doi: 10.1148/radiol.10100161. No abstract available. PMID 21273517
- [Background] Schoenhagen P, Nagel E. Noninvasive assessment of coronary artery disease anatomy, physiology, and clinical outcome. JACC Cardiovasc Imaging. 2011 Jan;4(1):62-4. doi: 10.1016/j.jcmg.2010.11.002. No abstract available. PMID 21232705
- [Result] Dewey M, Rief M, Martus P, Kendziora B, Feger S, Dreger H, Priem S, Knebel F, Bohm M, Schlattmann P, Hamm B, Schonenberger E, Laule M, Zimmermann E. Evaluation of computed tomography in patients with atypical angina or chest pain clinically referred for invasive coronary angiography: randomised controlled trial. BMJ. 2016 Oct 24;355:i5441. doi: 10.1136/bmj.i5441. PMID 27777234
- [Result] Bosserdt M, Feger S, Rief M, Preuss D, Ibes P, Martus P, Kofoed KF, Laule M, Perez I, Dewey M. Performing Computed Tomography Instead of Invasive Coronary Angiography: Sex Effects in Patients With Suspected CAD. JACC Cardiovasc Imaging. 2020 Mar;13(3):888-889. doi: 10.1016/j.jcmg.2019.10.014. Epub 2019 Dec 18. No abstract available. PMID 31864987
- [Derived] Bosserdt M, Mohamed M, Neumann K, Rieckmann N, Dreger H, Brodszky V, Hofer S, Reinhold T, Mielke AM, Dewey M. Cost-utility of computed tomography in patients with atypical chest pain clinically referred for invasive coronary angiography: randomised controlled trial. Eur Radiol. 2025 Nov;35(11):6719-6734. doi: 10.1007/s00330-025-11692-0. Epub 2025 May 24. PMID 40411549
- [Derived] Bosserdt M, Martus P, Tauber R, Dreger H, Dewey M, Schonenberger E; CAD-Man Study Group Investigators. Serum creatinine baseline fluctuation and acute kidney injury after intravenous or intra-arterial contrast agent administration-an intraindividual comparison as part of a randomized controlled trial. Nephrol Dial Transplant. 2022 May 25;37(6):1191-1194. doi: 10.1093/ndt/gfac013. No abstract available. PMID 35090035
- [Derived] Schonenberger E, Martus P, Bosserdt M, Zimmermann E, Tauber R, Laule M, Dewey M. Kidney Injury after Intravenous versus Intra-arterial Contrast Agent in Patients Suspected of Having Coronary Artery Disease: A Randomized Trial. Radiology. 2019 Sep;292(3):664-672. doi: 10.1148/radiol.2019182220. Epub 2019 Jul 2. PMID 31264950
- See also: CAD-Man results — http://www.bmj.com/content/355/bmj.i5441